CLINICAL TRIAL: NCT04888910
Title: Novel Inflammatory Markers in Different Phenotypes of Severe Asthma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Ilaria Puxeddu, Associate Professor, University of Pisa
Other Study IDs: NIMISA
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Asthma; Nasal Polyps
Keywords: asthma; eosinophils; neutrophils
MeSH Terms: conditions — Asthma; Nasal Polyps | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- asthma with nasal polyps: severe asthma with involvement of the upper airways (chronic rhinosinusitis with nasal polyps)
  Interventions: Other: observational
- severe asthma without nasal polyps: severe asthma without involvement of the upper airways
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — observation of biomarkers in different asthma groups

SUMMARY:
Asthma is a highly prevalent chronic airway inflammatory disease characterized by airway hyper-responsiveness, reversible airflow obstruction and increased mucus secretion, involving large and small airways. An emerging sub-phenotype of severe asthma is the late onset disease associated with nasal polyposis, a frequent co-morbidity that significantly impacts lung function and symptom control. On the basis of the infiltrate found in the sputum, asthma can be divided into four distinct phenotypes: eosinophilic, neutrophilic, mixed granulocytic and pauci-granulocytic. The majority of patients with eosinophilic asthma are sensitive to corticosteroids, and biological therapies targeting eosinophils (anti-Interleukin (IL)-5 and anti-IL5R) have been recently approved. However, it is known that some asthmatics, particularly those who have severe disease and are resistant to corticosteroids, have elevated neutrophil counts in the airway where they play a vital role in the exacerbation of the disease. However, the precise role of neutrophils in severe asthma and the mechanisms involved in neutrophil-induced tissue damage have not been clarified yet.

The hypothesis of the study is that neutrophils and eosinophils can contribute to the severity of asthma by changing their phenotypes according to the airway environment. Thus, a better understanding of the roles of neutrophils and eosinophils in severe asthma may lead to the identification of novel biomarkers and the development of new therapeutic approaches in different phenotypes of severe asthma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* age (18-65 years)
* Diagnosis of severe asthma according to the European Respiratory Society (ERS) and American Thoracic Society (ATS) definition, with and without nasal symptoms
* normal pulmonary function post-therapy (FEV1 post-bronchodilation: greater than 80% of the predicted value, with FEV1/ vital capacity (VC) > 88-89% - for males and females, respectively - of the predicted value)
* non reversible chronic airflow limitation (FEV1 post-bronchodilation: lower than 70% of the predicted value, with FEV1/VC < 88-89% of the predicted value)
* Signing of the informed consent

Exclusion Criteria:

* Referred Pregnancy
* Use of therapy with beta-blockers
* Smoking (current or within the previous 3 months)
* Negation to participate to the study
* Current upper and lower airways infectious diseases
* Current systemic infectious diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: severe asthmatic patients referred to the asthma clinic with or without upper airways involvement. Some of them are currently under biological therapies according to their grade of disease in addition to inhaled therapies.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
cell receptors | 2 years
  to identify neutrophil- and eosinophil-receptors in the airways of severe asthmatic patients with or without involvement of the upper airways
cell mediators | 2 years
  to identify soluble and matrix-derived mediators from neutrophils and eosinophils in the airways of severe asthmatic patients with or without involvement of the upper airways

CONTACTS AND LOCATIONS:
Locations (1):
- Pisa University, Pisa, Tuscany, Italy

REFERENCES:
- [Result] Wu W, Bleecker E, Moore W, Busse WW, Castro M, Chung KF, Calhoun WJ, Erzurum S, Gaston B, Israel E, Curran-Everett D, Wenzel SE. Unsupervised phenotyping of Severe Asthma Research Program participants using expanded lung data. J Allergy Clin Immunol. 2014 May;133(5):1280-8. doi: 10.1016/j.jaci.2013.11.042. Epub 2014 Feb 28. PMID 24589344
- [Result] Wenzel SE, Jayawardena S, Graham NM, Pirozzi G, Teper A. Severe asthma and asthma-chronic obstructive pulmonary disease syndrome - Authors' reply. Lancet. 2016 Dec 3;388(10061):2742. doi: 10.1016/S0140-6736(16)31720-2. Epub 2016 Dec 2. No abstract available. PMID 27924776
- [Result] Ray A, Kolls JK. Neutrophilic Inflammation in Asthma and Association with Disease Severity. Trends Immunol. 2017 Dec;38(12):942-954. doi: 10.1016/j.it.2017.07.003. Epub 2017 Aug 4. PMID 28784414